CLINICAL TRIAL: NCT04784078
Title: Randomized Comparison of Distal Radial Versus Conventional Radial Access for Coronary Angiography and Intervention
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Beijing Anzhen Hospital (Other)
Responsible Party: Principal Investigator, Yujie Zhou, Doctor, Beijing Anzhen Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DC radial
Record Dates: First submitted 2021-03-03; First posted 2021-03-05 (Actual); Last update posted 2021-04-13 (Actual); Status verified 2021-04

CONDITIONS: Coronary Disease
Keywords: Distal radial artery; Radial access
MeSH Terms: conditions — Coronary Disease | interventions — Methods

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- dTRA group (Experimental)
  Interventions: Procedure: Coronary Angiography and Intervention
- cTRA group (Active Comparator)
  Interventions: Procedure: Coronary Angiography and Intervention

INTERVENTIONS:
Procedure: Coronary Angiography and Intervention — Transradial access puncture site

SUMMARY:
Distal radial access (dTRA) represents a novel site for radial artery access in interventional cardiology, there is little data compare dTRA with conventional radial access (cTRA) in a randomized manner.

It aims to randomly compare between the new distal radial access via the snuffbox and the conventional radial access for percutaneous coronary intervention (PCI) and angioplasty procedures. The objectives of comparing both procedures are to analyze the frequency of complications in terms of occlusion, arterial spasm, hematoma, and to weigh accesses effectiveness in terms of time and attempts to puncture, crossover rate, procedure duration, hemostasis time.

Candidates for coronary angiography are being randomized into the interventional group to undergo the angiography through the distal radial artery as the access site, or the control group accessing through the radial artery. Procedural and post procedural outcomes and complications are being reported while patients are in hospital. All patients undergo doppler ultrasonography within 24 hours before and after the procedure, 4 weeks after procedure.

ELIGIBILITY:
Inclusion Criteria:

* Patient is over 18 years of age.
* Patient is undergoing diagnostic coronary angiography and/or PCI for the first time.
* Patient has provided written informed consent.
* Patient is willing to comply with all protocol-required evaluations during the hospitalization.

Exclusion Criteria:

* No palpable radial artery or distal radial artery.
* Radial artery used as a bridging vessel.
* Severe heart failure (NYHA class IV).
* Severe renal insufficiency ( SCr>443umol/L).
* Height over 185 cm.
* A ≥7F catheter may be required for operation.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 938 (Estimated)
Dates: Start 2021-04-10 (Estimated); Primary Completion 2021-12-31 (Estimated); Study Completion 2022-01-31 (Estimated)

PRIMARY OUTCOMES:
Radial artery occlusion | Within 24 hours after the procedure.
  Doppler Ultrasonography of the radial artery for occlusions along its course, in both groups. Incidence of radial artery occlusion as confirmed by absense of antegrade flow in vascular doppler ultrasound.

CONTACTS AND LOCATIONS:
Overall Officials: Yujie Zhou, Doctor, Study Chair — Beijing Anzhen Hospital

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Nikolakopoulos I, Vemmou E, Brilakis ES. Distal radial access for cardiac catheterization: When and how. Hellenic J Cardiol. 2020 Mar-Apr;61(2):110-111. doi: 10.1016/j.hjc.2020.06.001. Epub 2020 Jun 14. No abstract available. PMID 32553614
- [Result] Liontou C, Kontopodis E, Oikonomidis N, Maniotis C, Tassopoulos A, Tsiafoutis I, Lazaris E, Koutouzis M. Distal Radial Access: A Review Article. Cardiovasc Revasc Med. 2020 Mar;21(3):412-416. doi: 10.1016/j.carrev.2019.06.003. Epub 2019 Jun 8. PMID 31227393
- [Result] Sgueglia GA, Di Giorgio A, Gaspardone A, Babunashvili A. Anatomic Basis and Physiological Rationale of Distal Radial Artery Access for Percutaneous Coronary and Endovascular Procedures. JACC Cardiovasc Interv. 2018 Oct 22;11(20):2113-2119. doi: 10.1016/j.jcin.2018.04.045. PMID 30336816
- [Result] Koutouzis M, Kontopodis E, Tassopoulos A, Tsiafoutis I, Katsanou K, Rigatou A, Didagelos M, Andreou K, Lazaris E, Oikonomidis N, Maniotis C, Ziakas A. Distal Versus Traditional Radial Approach for Coronary Angiography. Cardiovasc Revasc Med. 2019 Aug;20(8):678-680. doi: 10.1016/j.carrev.2018.09.018. Epub 2018 Oct 2. PMID 30314833
- [Result] Xenogiannis I, Brilakis ES. Distal radial access at the anatomic snuffbox: The new standard for left radial access? Catheter Cardiovasc Interv. 2019 Nov 1;94(5):658-659. doi: 10.1002/ccd.28551. No abstract available. PMID 31675155